CLINICAL TRIAL: NCT02699190
Title: LeukoSEQ: Whole Genome Sequencing as a First-Line Diagnostic Tool for Leukodystrophies
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Adeline Vanderver, MD, Program Director, Leukodystrophy Center, Children's Hospital of Philadelphia
Other Study IDs: 16-013213
Record Dates: First submitted 2016-02-16; First posted 2016-03-04 (Estimated); Results first posted 2025-06-15 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Leukodystrophy; White Matter Disease; 4H Syndrome; Adrenoleukodystrophy; AMN; ALD; ALD (Adrenoleukodystrophy); X-linked Adrenoleukodystrophy; X-ALD; Adrenomyeloneuropathy; Aicardi Goutieres Syndrome; AGS; Alexander Disease; Alexanders Leukodystrophy; AxD; ADLD; Canavan Disease; CTX; Cerebrotendinous Xanthomatoses; Krabbe Disease; GALC Deficiency; Globoid Leukodystrophy; TUBB4A-Related Leukodystrophy; H-ABC - Hypomyelination, Atrophy of Basal Ganglia and Cerebellum; HBSL; HBSL - Hypomyelination, Brain Stem, Spinal Cord, Leg Spasticity; LBSL; Leukoencephalopathy With Brain Stem and Spinal Cord Involvement and High Lactate Syndrome (Disorder); Leukoencephalopathy With Brainstem and Spinal Cord Involvement and Lactate Elevation; ALSP; CSF1R Gene Mutation; HCC - Hypomyelination and Congenital Cataract; MLC1; Megalencephalic Leukoencephalopathy With Subcortical Cysts 1; MLD; Metachromatic Leukodystrophy; PMD; Pelizaeus-Merzbacher Disease; PLP1 Null Syndrome; PLP1 Gene Duplication | Blood or Tissue | Mutations; Pelizaeus-Merzbacher-Like Disease, 1; Peroxisomal Biogenesis Disorder; Zellweger Syndrome; Refsum Disease; Salla Disease; Sialic Storage Disease; Sjögren; Sjogren-Larsson Syndrome; Van Der Knapp Disease; Vanishing White Matter Disease; Charcot-Marie-Tooth; CMT; Mct8 (Slc16A2)-Specific Thyroid Hormone Cell Transporter Deficiency; Allan-Herndon-Dudley Syndrome; Cadasil; Cockayne Syndrome; Multiple Sulfatase Deficiency; Gangliosidoses; GM2 Gangliosidosis; BPAN; Labrune Syndrome; LCC; Mucopolysaccharidoses; TBCK-Related Intellectual Disability Syndrome
Keywords: Leukodystrophy; White Matter Disease; Whole Genome Sequencing; WGS
MeSH Terms: conditions — Leukoencephalopathies; Attention Deficit Disorder with Hyperactivity; Adrenoleukodystrophy; Aicardi-Goutieres syndrome; Alexander Disease; Alexanders leukodystrophy; Canavan Disease; Xanthomatosis, Cerebrotendinous; Leukodystrophy, Globoid Cell; Leukodystrophy, Hypomyelinating, 6; Leukoencephalopathy with Brainstem and Spinal Cord Involvement and Lactate Elevation; Leukodystrophy, Hypomyelinating, 5; Megalencephalic leukoencephalopathy with subcortical cysts; Leukodystrophy, Metachromatic; Pelizaeus-Merzbacher Disease; Leukodystrophy, Hypomyelinating, 2; Peroxisomal Disorders; Zellweger Syndrome; Refsum Disease; Sialic Acid Storage Disease; Sjogren's Syndrome; Sjogren-Larsson Syndrome; Charcot-Marie-Tooth Disease; Allan-Herndon-Dudley syndrome; CADASIL; Cockayne Syndrome; Multiple Sulfatase Deficiency Disease; Gangliosidoses; Gangliosidoses, GM2; Leukoencephalopathy Brain Calcifications and Cysts; Mucopolysaccharidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Study Cohort: This cohort comprises recently identified individuals for whom a clinical decision has been made to pursue whole genome sequencing (WGS) as a first-line diagnostic test. The cohort also includes each subject's biological parents.

SUMMARY:
Leukodystrophies, and other heritable disorders of the white matter of the brain, were previously resistant to genetic characterization, largely due to the extreme genetic heterogeneity of molecular causes. While recent work has demonstrated that whole genome sequencing (WGS), has the potential to dramatically increase diagnostic efficiency, significant questions remain around the impact on downstream clinical management approaches versus standard diagnostic approaches.

DETAILED DESCRIPTION:
Leukodystrophies are a group of approximately 30 genetic diseases that primarily affect the white matter of the brain, a complex structure composed of axons sheathed in myelin, a glial cell-derived lipid-rich membrane. Leukodystrophies are frequently characterized by early onset, spasticity and developmental delay, and are degenerative in nature. As a whole, leukodystrophies are relatively common (approximately 1 in 7000 births or almost twice as prevalent as Prader-Willi Syndrome, which has been far more extensively studied) with high associated health-care costs; however, more than half of the suspected leukodystrophies do not have a definitive diagnosis, and are generally classified as "leukodystrophies of unknown etiology". Even when a diagnosis is achieved, the diagnostic process lasts an average of eight years and results in test expenses in excess of $8,000 on average per patient, including the majority of patients who never achieve a diagnosis at all. These diagnostic challenges represent an urgent and unresolved gap in knowledge and disease characterization, as obtaining a definitive diagnosis is of paramount importance for leukodystrophy patients. The diagnostic workup begins with findings on cranial Magnetic Resonance Imaging (MRI) followed by sequential targeted genetic testing, however next generation sequencing (NGS) technologies offer the promise of rapid and more cost effective approaches.

Despite significant advances in diagnostic efficacy, there are still significant issues with respect to implementation of NGS in clinical settings. First, sample cohorts demonstrating diagnostic efficacy are generally small, retrospective, and susceptible to ascertainment bias, ultimately rendering them poor candidates for utility analyses (to determine how efficient a test is at producing a diagnosis). Second, historic sample cohorts have not been examined prospectively for information about impact on clinical management (whether the test results in different clinical monitoring, a change in medications, or alternate clinical interventions).

To address these issues, the study team conducted an investigation of patients with suspected leukodystrophies or other genetic disorders affecting the white matter of the brain at the time of initial confirmation of MRI abnormalities, with prospective collection of patients randomly received on a "first come, first served" basis from a network of expert clinical sites. Subjects were randomized to receive early (1 month) or late (6 months) WGS, with SoC clinical analyses conducted alongside WGS testing. An interim analysis performed in May 2018 assessed these study outcomes for a cohort of thirty-four (34) enrolled subjects. Two of these subjects were resolved before complete enrollment and were retained as controls. Nine subjects were stratified to the Immediate Arm, of which 5 (55.6%) were resolved by WGS and 4 (44.4%) were persistently unresolved. Of the 23 subjects randomized to the Delayed Arm, 14 (60.9%) were resolved by WGS and 5 (21.7%) by SoC, while the remaining 4 (17.4%) remained undiagnosed. The diagnostic efficacy of WGS in both arms was significant relative to SoC (p<0.005). The time to diagnosis was significantly shorter in the immediate WGS group (p<0.05). The overall diagnostic efficacy of the combination of WGS and SoC approaches was 26/34 (76.5%; 95% CI = 58.8% to 89.3%) over <4 months, greater than historical norms of <50% over more than 5 years.

The study now seeks to determine whether WGS results in changes to diagnostic status and clinical management in subjects affected by undiagnosed genetic disorders of the white matter of the brain. We anticipate that WGS will produce measurable downstream changes in diagnostic status and clinical management, as defined by disease-specific screening for complications or implementation of disease-specific therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Abnormalities of the white matter signal on neuroimaging (MRI) with T2 hyperintensity which must be diffuse or involve specific anatomical tracts consistent with a genetic diagnosis;
2. No pre-existing genetic diagnosis;
3. A clinical decision has been made to perform WGS;
4. Less than 18 years of age (exception for the affected sibling of the proband);
5. Availability of both biologic parents for blood sampling;
6. Availability of both biological parents to provide informed consent;
7. Concurrently enrolled in CHOP IRB 14-011236 (Myelin Disorders Biorepository Project)

Exclusion Criteria:

1. Candidates with acquired disorders, including infection, acute disseminated encephalomyelitis (ADEM), multiple sclerosis, vasculitis or toxic leukoencephalopathies;
2. Patients who have had previous genetic testing*, including WES or WGS;
3. Those with no third-party payer insurance, unable to receive standard of care diagnosis and therapeutic approaches;
4. Candidates who have already received a diagnosis.

   * Note: Karyotype or microarray testing that did not yield a definitive diagnosis should not be considered as an excluding factor.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We expect participants to be identified during their initial presentation and preliminary diagnostic workup. Leukodystrophies are heritable conditions that - with only few exceptions - are not gender-specific. We therefore expect males and females to be equally represented in the study population. The age of presentation is variable ranging from infancy to adulthood, though enrollment for the study is limited to individuals who have not yet reached the age of 18. All ethnicities are equally represented in these disorders, and we expect ethnicities to be represented based on US census data of population distribution.
Sampling Method: Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Vanderver, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) only available to principal investigator, co-investigators, and trial staff.

REFERENCES:
- [Background] Costello DJ, Eichler AF, Eichler FS. Leukodystrophies: classification, diagnosis, and treatment. Neurologist. 2009 Nov;15(6):319-28. doi: 10.1097/NRL.0b013e3181b287c8. PMID 19901710
- [Background] Bonkowsky JL, Nelson C, Kingston JL, Filloux FM, Mundorff MB, Srivastava R. The burden of inherited leukodystrophies in children. Neurology. 2010 Aug 24;75(8):718-25. doi: 10.1212/WNL.0b013e3181eee46b. Epub 2010 Jul 21. PMID 20660364
- [Background] Vanderver A, Hussey H, Schmidt JL, Pastor W, Hoffman HJ. Relative incidence of inherited white matter disorders in childhood to acquired pediatric demyelinating disorders. Semin Pediatr Neurol. 2012 Dec;19(4):219-23. doi: 10.1016/j.spen.2012.10.001. PMID 23245555
- [Background] Richards J, Korgenski EK, Srivastava R, Bonkowsky JL. Costs of the diagnostic odyssey in children with inherited leukodystrophies. Neurology. 2015 Sep 29;85(13):1167-70. doi: 10.1212/WNL.0000000000001974. Epub 2015 Aug 28. PMID 26320197
- [Background] Richards J, Korgenski EK, Taft RJ, Vanderver A, Bonkowsky JL. Targeted leukodystrophy diagnosis based on charges and yields for testing. Am J Med Genet A. 2015 Nov;167A(11):2541-3. doi: 10.1002/ajmg.a.37215. Epub 2015 Jul 16. PMID 26183797
- [Background] Bamshad MJ, Ng SB, Bigham AW, Tabor HK, Emond MJ, Nickerson DA, Shendure J. Exome sequencing as a tool for Mendelian disease gene discovery. Nat Rev Genet. 2011 Sep 27;12(11):745-55. doi: 10.1038/nrg3031. PMID 21946919
- [Background] Srivastava S, Cohen JS, Vernon H, Baranano K, McClellan R, Jamal L, Naidu S, Fatemi A. Clinical whole exome sequencing in child neurology practice. Ann Neurol. 2014 Oct;76(4):473-83. doi: 10.1002/ana.24251. Epub 2014 Aug 30. PMID 25131622
- [Background] Vanderver A, Simons C, Helman G, Crawford J, Wolf NI, Bernard G, Pizzino A, Schmidt JL, Takanohashi A, Miller D, Khouzam A, Rajan V, Ramos E, Chowdhury S, Hambuch T, Ru K, Baillie GJ, Grimmond SM, Caldovic L, Devaney J, Bloom M, Evans SH, Murphy JLP, McNeill N, Fogel BL; Leukodystrophy Study Group; Schiffmann R, van der Knaap MS, Taft RJ. Whole exome sequencing in patients with white matter abnormalities. Ann Neurol. 2016 Jun;79(6):1031-1037. doi: 10.1002/ana.24650. Epub 2016 May 9. PMID 27159321
- [Background] Schiffmann R, van der Knaap MS. Invited article: an MRI-based approach to the diagnosis of white matter disorders. Neurology. 2009 Feb 24;72(8):750-9. doi: 10.1212/01.wnl.0000343049.00540.c8. PMID 19237705
- [Derived] Vanderver A, Bernard G, Helman G, Sherbini O, Boeck R, Cohn J, Collins A, Demarest S, Dobbins K, Emrick L, Fraser JL, Masser-Frye D, Hayward J, Karmarkar S, Keller S, Mirrop S, Mitchell W, Pathak S, Sherr E, van Haren K, Waters E, Wilson JL, Zhorne L, Schiffmann R, van der Knaap MS, Pizzino A, Dubbs H, Shults J, Simons C, Taft RJ; LeukoSEQ Workgroup. Randomized Clinical Trial of First-Line Genome Sequencing in Pediatric White Matter Disorders. Ann Neurol. 2020 Aug;88(2):264-273. doi: 10.1002/ana.25757. Epub 2020 Jun 9. PMID 32342562
- See also: CHOP Leukodystrophy Center Research Portal — https://www.chop.edu/centers-programs/leukodystrophy-center/research

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospective Study Cohort
Started | 236
Affected Patients | 80
Biological Parents | 156
Completed | 236
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline data was only obtained from affected patients. Biological parents' medical records were collected and reviewed to verify whether the affected patient's genetic variant was pathogenic. Therefore, the baseline analysis population includes the 80 enrolled affected patients and excludes the 156 enrolled biological parents.
Arm/Group | Prospective Study Cohort
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 80
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 60
  More than one race | 4
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Changes in Diagnosis Status (Resulting From WGS)
Description: The primary objective of this study is to evaluate changes in diagnostic status in the study cohort for patients who received Whole Genome Sequencing (WGS) as part of clinical care. Differences in diagnostic status will be measured at disclosure of initial results or disclosure of reanalyzed results.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Study Cohort
Number analyzed (Participants) | 80
Participants | 45

2. Secondary Outcome: Changes in Clinical Management (Resulting From WGS)
Description: The secondary objective of this study is to evaluate changes in clinical care in subjects who received a diagnosis through Whole Genome Sequencing (WGS). Differences in clinical care will be evaluated 1 year following disclosure of results.
Time Frame: 12 months
Population: There were 45/80 participants with diagnostic results and 38 of these subjects had sufficient medical records for 1-year post-Genomic Sequencing (GS) review.
  The numbers included below (37, 35 and 8) overlap: one participant could be part of the 3 different rows counts.
Measure: Number; unit: participants
Arm/Group | Prospective Study Cohort
Number analyzed (Participants) | 38
participants
  Referred to specialists providers for disease monitoring | 37
  Received additional targeted screening | 35
  Eligible for disease modifying treatment | 8

ADVERSE EVENTS:
Time Frame: This study is observational and considered to involve no greater than minimal risk. The primary risk of study participation involves breach of confidentiality due to collection, analysis, and/or retention of Personal Health Information (PHI) from subject medical records. Adverse events were therefore not expected and not collected.
Description: Due to the nature of the study, adverse events were not expected and not collected.
Arm/Group | Prospective Study Cohort
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT02699190/Prot_SAP_001.pdf
  • Informed Consent Form (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT02699190/ICF_002.pdf